CLINICAL TRIAL: NCT01708265
Title: Dutch AMR; Early Mitral Valve Repair Versus Watchful Waiting in Asymptomatic Patients With Severe Organic Mitral Regurgitation; a Multicenter, Randomised Trial.
Brief Title: The Dutch Asymptomatic Mitral Regurgitation Trial
Acronym: Dutch AMR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low inclusion rate
Sponsor: UMC Utrecht (Other)
Collaborators: Leiden University Medical Center (Other); The Interuniversity Cardiology Institute of the Netherlands (Other Government); WCN, Dutch Network for Cardiovascular Research (Unknown)
Responsible Party: Principal Investigator, S.A.J. Chamuleau, MD, PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL39851.041.12.
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Heart; Disease, Mitral(Valve); Diseases of Mitral Valve; Mitral Valve Insufficiency
Keywords: Mitral Valve Insufficiency; Mitral Valve Regurgitation; Asymptomatic Mitral Valve Regurgitation; Asymptomatic Mitral Valve Insufficiency; Mitral Valve Repair; Watchful Waiting
MeSH Terms: conditions — Disease; Mitral Valve Insufficiency | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early mitral valve repair (Active Comparator): Early mitral valve repair
  Interventions: Procedure: Early mitral valve repair
- Watchful waiting (Active Comparator): Watchful waiting
  Interventions: Other: Watchful waiting

INTERVENTIONS:
Other: Watchful waiting — In case of watchful waiting a conservative treatment is performed, based on close monitoring of the patient for clear signs of deterioration that triggers facilitated surgery before left ventricular dysfunction is present.
  Arms: Watchful waiting
Procedure: Early mitral valve repair — Patients in the group of early mitral valve repair will be operated by way of routine mitral valve repair procedures in specialized centres.
  Arms: Early mitral valve repair

SUMMARY:
The purpose of this study is to compare early mitral valve repair versus a watchful waiting strategy in asymptomatic patients with severe organic mitral valve regurgitation and preserved left ventricular function.

DETAILED DESCRIPTION:
Severe asymptomatic organic mitral valve (MV) regurgitation with preserved left ventricular (LV) function is a challenging clinical entity as data on the recommended treatment strategy for these patients are scarce and conflicting, which is reflected in current guidelines. European guidelines advocate a more conservative strategy i.e. watchful waiting, with yearly echocardiography, whilst American guidelines are more in favour of early surgery to reconstruct the MV, i.e. MV repair (in contrast to MV replacement) in order to prevent future LV dysfunction and complaints.

A number of non-randomised trials show a favourable outcome of early surgery and the early surgery strategy has shown to be associated with improved long-term survival, decreased cardiac mortality and decreased morbidity compared with the conservative management [citations 1-3]. On the other hand, non-randomised trials describe also that a conservative strategy (i.e. watchful waiting) can be safely accomplished. If facilitated surgery is performed in this population it has proven to be eventually associated with good perioperative and postoperative outcome in 50% of the patients at 10 years when careful follow-up is being carried out [citation 4]. Non-randomised trials inherently have a number of drawbacks. A randomised trial comparing both strategies and objectivising the best treatment strategy has never been performed.

The Dutch AMR (Asymptomatic Mitral Regurgitation) trial is a multicenter, prospective, randomised trial comparing early MV repair versus watchful waiting in asymptomatic patients with severe organic MV regurgitation and preserved LV function [citation 5, 6].

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic
* Severe organic mitral valve regurgitation.
* Preserved left ventricular function (left ventricular ejection fraction >60% and left ventricular end-systolic dimension ≤45 mm)
* The likelihood of MV repair should be more than 90% determined by the local heart team with a cardiologist and cardiothoracic surgeon

Exclusion Criteria:

* Pulmonary hypertension (>50 mmHg at rest)
* Atrial fibrillation
* Physical inability as determined by the heart team to undergo surgery
* Other life-threatening morbidity
* Higher expected surgical risks in advance, according to the dedicated heart team
* Moderate to severe kidney disease (eGFR less than 30 mL/min)
* Flail leaflet together with a left ventricular end systolic diameter (LVESD) >40 mm

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02; Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint: cardiovascular mortality, congestive heart failure and hospitalization for nonfatal cardiovascular events | Min. 5 years
  The primary outcome is defined as 'time to first event'. It concerns time to first event of the composite endpoint of cardiovascular mortality, congestive heart failure, non-fatal cardiovascular events requiring hospitalization, defined as: stroke/cerebrovascular accident (CVA), atrial fibrillation (permanent or requiring hospitalization) and/or reoperation after elective MV surgery.

SECONDARY OUTCOMES:
Cardiovascular mortality | Min. 5 years
  Secondary outcome measures are the separate components of the composite primary endpoint: cardiovascular mortality, congestive heart failure, hospitalization for nonfatal cardiovascular events (stroke/cerebrovascular accident (CVA), AF (permanent or requiring hospitalization) and reoperation after elective MV surgery).
Congestive heart failure | Min. 5 years
  Secondary outcome measures are the separate components of the composite primary endpoint: cardiovascular mortality, congestive heart failure, hospitalization for nonfatal cardiovascular events (stroke/cerebrovascular accident (CVA), AF (permanent or requiring hospitalization) and reoperation after elective MV surgery).
Hospitalization for nonfatal cardiovascular events | Min. 5 years
  Secondary outcome measures are the separate components of the composite primary endpoint: cardiovascular mortality, congestive heart failure, hospitalization for nonfatal cardiovascular events (stroke/cerebrovascular accident (CVA), AF (permanent or requiring hospitalization) and reoperation after elective MV surgery).
All-cause mortality | Min. 5 years
  Secondary outcome measures the incidence of all-cause mortality at a minimum of 5 years.
Costs and effectiveness | Min. 5 years
  Secondary outcome measures total direct and indirect costs and cost-effectiveness at a minimum of 5 years.
Health-related quality of life | Min. 5 years
  Secondary outcome measures health-related quality of life at a minimum of 5 years.
Echocardiographic parameters | Min. 5 years
  Secondary outcome measures echocardiographic parameters at a minimum of 5 years.
CMR parameters | Min. 5 years.
  Secondary outcome measures Cardiovascular Magnetic Resonance imaging (CMR) parameters at a minimum of 5 years.
Paroxysmal atrial fibrillation | Min. 5 years
  Secondary outcome measures the incidence of paroxysmal atrial fibrillation at a minimum of 5 years.
Exercise test parameters | Min. 5 years.
  Secondary outcome measures exercise test parameters at a minimum of 5 years.
BNP | Min. 5 years
  Secondary outcome measures brain natriuretic peptide (BNP) plasma levels at a minimum of 5 years.
Myocardial infarction | Min. 5 years
  Secondary outcome measures the incidence of myocardial infarction at a minimum of 5 years.
Pacemaker implantation | Min. 5 years
  Secondary outcome measures the incidence of pacemaker implantation at a minimum of 5 years.
Transient ischemic attack | Min. 5 years
  Secondary outcome measures the incidence of transient ischemic attack (TIA) at a minimum of 5 years.
Pulmonary embolism | Min. 5 years
  Secondary outcome measures the incidence of pulmonary embolism at a minimum of 5 years.

OTHER OUTCOMES:
Surgery complication rate | Min. 5 years
  The complication rate in the mitral valve surgery group (e.g. re-operation for bleeding, pneumonia, residual or recurrent mitral valve regurgitation) will be determined at a minimum of 5 years.
Rate for the need of facilitated surgery | Min. 5 years
  Rate for the need of facilitated surgery in the watchful waiting group will be determined at a minimum of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Steven AJ Chamuleau, MD, PhD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht); Jolanda Kluin, MD, PhD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht); Robert JM Klautz, Prof. MD PhD, Principal Investigator — Leiden University Medical Center (LUMC Leiden)
Locations (4):
- Netherlands (4):
  - Leiden University Medical Center, Leiden, South Holland
  - University Medical Center Utrecht (UMC Utrecht), Utrecht, Utrecht
  - Amsterdam Medisch Centrum, Amsterdam
  - Amphia Hospital, Breda

REFERENCES:
- [Background] Ling LH, Enriquez-Sarano M, Seward JB, Orszulak TA, Schaff HV, Bailey KR, Tajik AJ, Frye RL. Early surgery in patients with mitral regurgitation due to flail leaflets: a long-term outcome study. Circulation. 1997 Sep 16;96(6):1819-25. doi: 10.1161/01.cir.96.6.1819. PMID 9323067
- [Background] Enriquez-Sarano M, Avierinos JF, Messika-Zeitoun D, Detaint D, Capps M, Nkomo V, Scott C, Schaff HV, Tajik AJ. Quantitative determinants of the outcome of asymptomatic mitral regurgitation. N Engl J Med. 2005 Mar 3;352(9):875-83. doi: 10.1056/NEJMoa041451. PMID 15745978
- [Background] Chenot F, Montant P, Vancraeynest D, Pasquet A, Gerber B, Noirhomme PH, El Khoury G, Vanoverschelde JL. Long-term clinical outcome of mitral valve repair in asymptomatic severe mitral regurgitation. Eur J Cardiothorac Surg. 2009 Sep;36(3):539-45. doi: 10.1016/j.ejcts.2009.02.063. Epub 2009 Jul 25. PMID 19632855
- [Background] Rosenhek R, Rader F, Klaar U, Gabriel H, Krejc M, Kalbeck D, Schemper M, Maurer G, Baumgartner H. Outcome of watchful waiting in asymptomatic severe mitral regurgitation. Circulation. 2006 May 9;113(18):2238-44. doi: 10.1161/CIRCULATIONAHA.105.599175. Epub 2006 May 1. PMID 16651470
- [Background] Tietge WJ, de Heer LM, van Hessen MW, Jansen R, Bots ML, van Gilst W, Schalij M, Klautz RJ, Van den Brink RB, Van Herwerden LA, Doevendans PA, Chamuleau SA, Kluin J. Early mitral valve repair versus watchful waiting in patients with severe asymptomatic organic mitral regurgitation; rationale and design of the Dutch AMR trial, a multicenter, randomised trial. Neth Heart J. 2012 Mar;20(3):94-101. doi: 10.1007/s12471-012-0249-y. PMID 22354529
- [Background] Jansen R, Kluin J, Chamuleau SA. Research versus clinical practice in asymptomatic patients with severe organic mitral regurgitation and preserved LV function. J Am Coll Cardiol. 2014 Oct 14;64(15):1639-40. doi: 10.1016/j.jacc.2014.07.964. No abstract available. PMID 25301470
- See also: Dutch AMR study homepage — http://dutchamr.nl/